CLINICAL TRIAL: NCT00381732
Title: A Randomized, Double-Blind, Parallel, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Tadalafil (2.5mg and 5mg) Administered Once Daily to Men With Erectile Dysfunction
Brief Title: A Study to Evaluate the Efficacy and Safety of 2.5mg and 5mg Tadalafil Given Once a Day to Men With Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7019; H6D-MC-LVFP
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2007-11

CONDITIONS: Erectile Dysfunction
Keywords: Impotence; erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): placebo tablet
  Interventions: Drug: placebo
- 2 (Active Comparator): 2.5 mg tadalafil tablet
  Interventions: Drug: tadalafil
- 3 (Active Comparator): 5 mg tadalafil tablet
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 2.5 mg or 5 mg tadalafil tablet taken by mouth once a day for 24 weeks. Followed by an open label extension where all patients receive 5 mg doses.
  Other Names: LY450190; Cialis; IC351
  Arms: 2; 3
Drug: placebo — Placebo tablet taken by mouth once a day for 24 weeks. Placebo patient will receive 5 mg tadalafil tablet during the open label extension.
  Arms: 1

SUMMARY:
This is a multicenter, randomized, double blind, placebo-controlled, parallel design study to evaluate the efficacy and safety of 2.5mg and 5mg tadalafil taken once daily in men with erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Men with erectile dysfunction
* At least 18 years of age

Exclusion Criteria:

* Certain chronic medical conditions including cardiac disease, congestive heart failure, kidney or liver disease, cancer and HIV
* A history of certain impotence disorders
* History of specified pelvic surgery
* Any significant genital abnormality identified at the start of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2003-10; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Changes in erectile function measured at baseline and after 6 months of treatment with 2.5mg and 5mg tadalafil; assessment of safety after 1 and 2 years of therapy with 5mg tadalafil. | 24-128 weeks

SECONDARY OUTCOMES:
Changes in additional aspects of erectile function after 3 and 6 months of treatment; assessment of the pharmacokinetics of tadalafil 2.5mg and 5mg. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bothell, Washington, United States

REFERENCES:
- [Derived] Porst H, Gacci M, Buttner H, Henneges C, Boess F. Tadalafil once daily in men with erectile dysfunction: an integrated analysis of data obtained from 1913 patients from six randomized, double-blind, placebo-controlled, clinical studies. Eur Urol. 2014 Feb;65(2):455-64. doi: 10.1016/j.eururo.2013.09.037. Epub 2013 Oct 2. PMID 24119319
- [Derived] Shabsigh R, Seftel AD, Kim ED, Ni X, Burns PR. Efficacy and safety of once-daily tadalafil in men with erectile dysfunction who reported no successful intercourse attempts at baseline. J Sex Med. 2013 Mar;10(3):844-56. doi: 10.1111/j.1743-6109.2012.02898.x. Epub 2012 Oct 4. PMID 23035781
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com